CLINICAL TRIAL: NCT05403879
Title: Modified Hook Wiring Technique for Greater Tuberosity Fractures, a Prospective Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Amr Elshahhat, MD., lecturer of orthopedics, Mansoura University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R.22.03.1644
Record Dates: First submitted 2022-05-31; First posted 2022-06-03 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2024-01

CONDITIONS: Greater Tuberosity Fractures
MeSH Terms: conditions — Shoulder Fractures

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- cases undergoing fixation of fractured greater tuberosity (Experimental)
  Interventions: Procedure: fixation of greater tuberosity fractures

INTERVENTIONS:
Procedure: fixation of greater tuberosity fractures — deltopectoral approach for shoulder, then open reduction and fixation of displaced greater tuberosity fractures using hooked Kirshner wires

SUMMARY:
the purpose of this study is to assess functional and radiological outcome of open reduction and internal fixation of isolated displaced greater tuberosity fractures (more than 5mm displacement) in adults advocating modified hook wiring with a follow-up period of one year.

DETAILED DESCRIPTION:
after being informed about the study and potential risks, all enrolled cases giving informed consent will undergo fixation of their fractured greater tuberosity, then physiotherapy. patients will be followed up till full union, clinical and radiological follow up for at least one year utilizing approved clinical scores and radiological criteria for healing. any complication will be recorded.

ELIGIBILITY:
Inclusion Criteria:

Patients presented and admitted at Mansoura Trauma, emergency hospital affiliated to Mansoura university, with acute isolated displaced GT fractures ( more than 5mm displacement), with/without glenohumeral dislocations, with age between 18years to 50 years.

Exclusion Criteria:

1. Skeletally immature patients (less than 18 years), age more than 50 years.
2. Open and pathological fractures
3. Associated proximal humeral fractures
4. History of previous GH dislocations
5. History of previous shoulder injuries or surgeries

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2022-03-23 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
functional outcome using American Shoulder and Elbow Surgeons (ASES) Standardized Shoulder Assessment score | at least one year follow up
  postoperative assessing pain, range of motion, function of shoulder. Scores range from 0 to 100 with a score of 0 indicating a worse shoulder condition and 100 indicating a better shoulder condition

SECONDARY OUTCOMES:
healing time | anticipated 2-4 months
  estimate time till radiological healing on follow-up radiographs

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura university hospital, Al Mansurah, Dakahlia Governorate, Egypt

REFERENCES:
- [Derived] Elshahhat A, Nour K. Modified Hook Wiring Technique for Greater Tuberosity Fractures: A Prospective Study. Acta Orthop Belg. 2025 Jun;91(2):209-220. doi: 10.52628/91.2.13849. PMID 40878734